CLINICAL TRIAL: NCT00781144
Title: The Effect of Experience and Gender on the Palpatory Forces Exerted by Novice and Experienced Osteopaths in Australia
Brief Title: Determination of Forces Used in Palpatory Diagnosis
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Responsible Party: Yasmin Qureshi, Nova Southeastern University
Other Study IDs: HPD-OST06030201X
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: first year osteopathic students
- 2: fourth and fifth year osteopathic students
- 3: experienced osteopathic clinicians

SUMMARY:
In this study, we are experimentally investigating the assessment of forces used by skilled clinicians and beginning practitioners in palpatory techniques. The study will assess pressure used during palpatory diagnosis of the paraspinal region.

DETAILED DESCRIPTION:
The study will assess pressure used during palpatory diagnosis of the paraspinal region. The research hypothesis is that both experience and gender will affect the amount of pressure exerted with diagnostic springing. The data will be valuable in characterizing practice parameters of novice and skilled osteopathic clinicians in palpation and will provide data on skill maturation from novice to experienced clinician. It will also allow far more precise teaching of these skills to students, who can use the transducers to determine how much pressure they are using compared to skilled clinicians. For measuring the palpatory forces, a thin film pressure transducer will be used in the hand of the clinician. Data will be collected on a portable computer via an analog to digital interface.

ELIGIBILITY:
Inclusion Criteria:

* osteopathic student first year or senior or experienced osteopathic clinician

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: first year osteopathic students, fourth and fifth year osteopathic students and experienced osteopathic clinicians
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
palpatory force exerted with PA springing | 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Qureshi, MHS. MPT, Principal Investigator — Nova Southeastern University, Victoria University
Locations (2):
- Nova Southeastern University, Fort Lauderdale, Florida, United States
- Victoria University, Melbourne, Victoria, Australia